CLINICAL TRIAL: NCT05766878
Title: The Rehabilitation of Atrophic Jaws Using Short Implants With Different Surface Characteristics: Multicentric RCT
Brief Title: The Rehabilitation of Atrophic Jaws Using Short Implants With Different Surface Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Collaborators: Universita degli Studi di Genova (Other); University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Khrystyna Zhurakivska, Researcher, University of Foggia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SHORT_1
Record Dates: First submitted 2023-02-10; First posted 2023-03-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Peri-Implantation Loss; Periodontal Bone Loss; Periimplantitis; Gingival Inflammation; Implant Complication; Osseointegration Failure of Dental Implant
Keywords: short implants; surface treatment
MeSH Terms: conditions — Alveolar Bone Loss; Peri-Implantitis; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- machined collar (Active Comparator): The arm will be constituted by healthy people, that need to be rehabilitated by dental implant placement.
  A short implant (length 6mm; diameter 4.3) will be inserted in an edentulous site. The implant will present a surface treated with double acid etching and traditional machined collar. A definitive transgingival standard machined abutment will be immediately screwed. Four months later, prosthetic procedures will start.
  Interventions: Device: implants placement
- anodized collar (Experimental): The arm will be constituted by healthy people, that need to be rehabilitated by dental implant placement.
  A short implant (length 6mm; diameter 4.3) will be inserted in an edentulous site. The implant will present a surface treated with double acid etching and anodized collar. A definitive transgingival anodized abutment will be immediately screwed. Four months later, prosthetic procedures will start.
  Interventions: Device: implants placement

INTERVENTIONS:
Device: implants placement — The intervention will consist of placement of two types of short implants (one with traditional machined collar and one with anodized collar). After their healing period, the prosthetic rehabilitation will be made.

SUMMARY:
The aim of the research is to evaluate the clinical outcome of short dental implants, characterized by a new macro-structural design and inserted in the upper or lower jaw in patients with reduced bone volume. The clinical outcomes will be compared for different surface treatments of implant neck and those of prosthetic components.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients, with edentulous maxillary or mandibular ridge, requiring rehabilitation with two adjacent implants;
* at least 6 month after extraction;

Exclusion Criteria:

* post-extractive implants;
* sites requiring bone regeneration or maxillary sinus lift;
* general health problems that contraindicate implant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Marginal Bone remodeling around the implant | 0-4-12 months after implant placement
  The marginal bone remodeling will be evaluated by Radiographic examination. Periapical radiographs will be performed using paralleling technique with a Rinn-type positioner, customized for each patient at implant placement (T0), prosthetic restoration delivery (T1), and after 12 months (T2).Peri-implant bone levels will be measured at each time point as the linear distance (in mm) between implant platform and bone crest at mesial and distal aspects of each implant. A positive value will be assigned if the bone crest is coronal to the implant platform, whereas a negative value will be assigned if the first bone-to implant contact is apical to the implant platform. All measurements will be performed by two examiners, using measuring software (Image J). Each measurement will be performed three times at three different points.

SECONDARY OUTCOMES:
Periodontal indexes: Probing Depth | The measurements will be performed at 4 (T1) and 12 (T2) months after implant placement.
  Probing Depth (PD) will be calculated as the distance (in mm) from the gingival peri-implant margin to the bottom of the peri-implant pocket.
Implant Stability evaluation | 0-4 months.
  Primary and secondary implant stability will be measured with resonance frequency analysis (RFA) and subsequently expressed as an implant stability quotient (ISQ). The Implant stability will be measured immediately after placement (T0) and at 4 months (T1) after placement, when the osseointegration is supposed to take place.
Bleeding on Probing | The measurements will be performed at 4 (T1) and 12 (T2) months after implant placement.
  Bleeding on probing (BoP) will be scored dichotomously (Yes/No). The probing will be performed on 6 sites around the implant (3 buccal and 3 palatal/lingual) and appearance of blood will be registered (Yes). The final score will be expressed as number of bleeding sites/total of probed sites (%)
Suppuration on probing | The measurements will be performed at 4 (T1) and 12 (T2) months after implant placement.
  Suppuration on probing (SUP) will be scored dichotomously (Yes/No). The probing will be performed on 6 sites around the implant (3 buccal and 3 palatal/lingual) and appearance of pus or purulent exudate will be registered (Yes). The final score will be expressed as number of suppurative sites/total of probed sites (%)
Plaque index of peri-implant tissues | The measurements will be performed at 4 (T1) and 12 (T2) months after implant placement.
  Plaque Index (PI) will be calculated by assigning a binary score to each surface (1= plaque present, 0 = plaque absent).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Troiano, DDS, PhD, Principal Investigator — University of Foggia; Francesco Pera, DDS, PhD, Study Chair — University of Turin, Italy
Locations (3):
- Italy (3):
  - Clinica Odontoiatrica, University of Foggia, Foggia
  - University of Genoa, Genova
  - University of Turin, Torino

IPD SHARING:
Plan to Share IPD: No
The data, in compliance with the privacy protection rules, will be shared upon request.

REFERENCES:
- [Derived] Longhi B, Pera F, Menini M, Bagnasco F, Pesce P, Caroprese M, Troiano G, Zhurakivska K. The Influence of Implant Surface Modification on Marginal Bone Loss and Periodontal Health: A Cross-Over Randomized Clinical Trial. Int J Dent. 2025 Sep 28;2025:8889144. doi: 10.1155/ijod/8889144. eCollection 2025. PMID 41059354